CLINICAL TRIAL: NCT06121063
Title: The Efficacy and Safety of a CCT-102 Regimen or Expectant Management in the Treatment of First Trimester Pregnancy Loss
Brief Title: CCT-102 or Expectant Management in Delayed Pregnancy Loss
Acronym: MERMAID
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Conceptra Biosciences, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PRT-CO-CCT-102.001
Record Dates: First submitted 2023-11-02; First posted 2023-11-07 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Early Pregnancy Loss, Delayed Pregnancy Loss
MeSH Terms: conditions — Abortion, Spontaneous

STUDY DESIGN:
Intervention Model Description: Open, label, multi-center, randomized study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- CCT-102 Regimen (Active Comparator): CCT-102 A/B regimen
  Interventions: Combination Product: CCT-102 A and CCT-102 B
- Expectant management (No Intervention): Non-treatment, 'waitful watching'

INTERVENTIONS:
Combination Product: CCT-102 A and CCT-102 B — 2 day oral regimen
  Arms: CCT-102 Regimen

SUMMARY:
A Phase 3, multi-center clinical trial of a CCT-102 regimen or expectant management to promote uterine evacuation in first trimester non-progressing Delayed Pregnancy Loss (DPL).

DETAILED DESCRIPTION:
This is a Phase 3, open-label, multi-center study to assess the efficacy of a CCT-102 regimen for uterine evacuation in first trimester delayed pregnancy loss (DPL). Eligible study participants will have ultrasound documented DPL with estimated gestational age 10 weeks or less.

DPL is defined as arrest of embryonic or fetal development, in first trimester, where the cervix is closed and there is no or only slight bleeding. This includes: 1) anembryonic pregnancy, and 2) embryonic demise. Expectant management, which is an accepted treatment protocol recognized in 2018 ACOG Practice Bulletin on Early Pregnancy Loss (ACOG, 2018), consists of patient monitoring with no additional treatment.

Eligible participants will choose between the investigational product or expectant management on Day 1. They will be evaluated for the primary endpoint (resolution of DPL) on Study Day 7. All participants will be followed to Day 28.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 to 50
2. Ability to provide informed consent
3. Hemodynamically stable
4. Closed cervical os
5. If fetus exists, clinical observation indicates gestation is no more than 10 weeks
6. Diagnosis of delayed pregnancy loss, confirmed by ultrasound, based on:

   1. Embryonic demise: no embryonic cardiac activity when embryo measures 7 mm or greater; OR,
   2. Anembryonic pregnancy: mean gestational sac diameter of 25 mm or greater, with no detectable embryo.

Exclusion Criteria:

1. Unwillingness or inability to comply with the study protocol and visit schedule
2. Diagnosis of an incomplete or inevitable abortion including more than slight bleeding at enrollment and/or open os within the prior week.
3. Confirmed or suspected ectopic pregnancy or undiagnosed adnexal mass
4. Hemoglobin <10 g/dL
5. Coagulation disorder, inherited porphyrias, and/or current anticoagulants use
6. Chronic adrenal failure
7. Concurrent chronic corticosteroid therapy
8. History of trophoblastic disease
9. Current presence of an IUD
10. History of allergy or contraindications to the use to mifepristone, misoprostol, or other prostaglandins
11. Any condition that, in the opinion of the investigator, makes the patient unsuitable for study entry
12. Any other current medical condition that jeopardizes the patient's ability to safely participate in the trial

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 183 (Actual)
Dates: Start 2023-07-21 (Actual); Primary Completion 2025-05-15 (Actual); Study Completion 2025-07-30 (Actual)

PRIMARY OUTCOMES:
Resolution of pregnancy loss | 7 Days
  Evacuation of delayed pregnancy loss within 7 days (up to and including Day 7), confirmed by ultrasound.

CONTACTS AND LOCATIONS:
Locations (15):
- United States (15):
  - Noble Clinical Research, Tucson, Arizona
  - Amicis Research Center, LLC, San Fernando, California
  - Emerald Coast Obstetrics and Gynecology, Panama City, Florida
  - Cypress Medical Research Center, Wichita, Kansas
  - Sinai Hospital of Baltimore, Baltimore, Maryland
  - Las Vegas Clinical Trials, Las Vegas, Nevada
  - Columbia University Irving Medical Center, New York, New York
  - Montefiore Medical Center, The Bronx, New York
  - Eastern Carolina Women's Center, PA, New Bern, North Carolina
  - Lyndhurst Clin Research, Winston-Salem, North Carolina
  - Penn State Hershey Obstetrics and Gynecology, Hershey, Pennsylvania
  - The University of Texas Medical Branch at Galveston, Galveston, Texas
  - Maximos Obstetrics & Gynecology, League City, Texas
  - Prime Clinical Research - Lewisville North Valley, Lewisville, Texas
  - Tidewater Clinical Research, Virginia Beach, Virginia

IPD SHARING:
Plan to Share IPD: No